CLINICAL TRIAL: NCT02899637
Title: Effects of High-Frequency Transcranial Magnetic Stimulation on Functional Performance of Subjects With Incomplete Spinal Cord Injury: Study Protocol for a Randomized Controlled Trial
Brief Title: Effects of Transcranial Magnetic Stimulation in Incomplete Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade Estadual da Paraiba (Other)
Responsible Party: Principal Investigator, Fernando Henrique Magalhães, Associate Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18753713.0.0000.5187
Record Dates: First submitted 2016-08-25; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Spinal Cord Injury
Keywords: Incomplete Spinal Cord Injury; Rehabilitation; Non-invasive brain stimulation; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spinal Cord Injury (Active Group) (Experimental): Active high-frequency Transcranial Magnetic Stimulation
  Interventions: Device: Active high-frequency Transcranial Magnetic Stimulation
- Spinal Cord Injury (Control group) (Sham Comparator): Sham high-frequency Transcranial Magnetic Stimulation
  Interventions: Device: Sham high-frequency Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Active high-frequency Transcranial Magnetic Stimulation — Active intervention, 5Hz on the lower limbs area of the motor cortex, during one week
  Arms: Spinal Cord Injury (Active Group)
Device: Sham high-frequency Transcranial Magnetic Stimulation — Sham intervention, 5Hz on the lower limbs area of the motor cortex, during one week
  Arms: Spinal Cord Injury (Control group)

SUMMARY:
The main objective is to conduct a study protocol to investigate the effects of repetitive Transcranial Magnetic Stimulation (rTMS) on sensory and motor performance of individuals with incomplete spinal cord injury (iSCI) . A double-blind randomized sham-controlled trial of patients with iSCI will be conducted.

DETAILED DESCRIPTION:
Effective rehabilitation programs for individuals with incomplete spinal cord injury (iSCI) are required either in the acute or in the post-acute care. Rehabilitation techniques based on protocols that selectively stimulate specific pathways along the central nervous system have been considered effective in enhancing neurologic recovery thereby improving functional abilities. The rationale relies on the assumption that the stimulation of the corticospinal tract, primary motor cortex, and spinal cord might induce neuronal reorganization of structures that are largely involved in the control of voluntary movements. In this line of reasoning, protocols involving repetitive transcranial magnetic stimulation (rTMS) have been found effective in enhancing corticospinal synaptic transmission, attenuating neuropathic pain, improving spasticity and sensorimotor function after iSCI. However, controversial findings have also been reported, as other studies showed unaltered central pain, as well as cortical excitability and sensorimotor function. The lack of consistent results is probably associated with differences in stimulation parameters, number of sessions, site of stimulation, chronicity and levels of injury, and outcome measurements of the previous studies. Thus, it is clear that there are remaining gaps in our knowledge and the development of new studies, preferably prospective fully double-blind placebo-controlled trials, is necessary to complement the current knowledge about the effects of rTMS in patients with iSCI.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of iSCI with nonprogressive etiology
* Clinical stability
* Aged between 18-60 years old
* Score equal to 24 in the Mini-Mental State Examination
* No electroencephalography alterations
* Absence of depression assessed by Hamilton Depression Scale
* Currently receiving inpatient rehabilitation in Physiotherapy Health Center of University of the State of Paraiba, Brazil.

Exclusion Criteria:

* Have metal prosthesis in some part of the body
* Use cardiac pacemaker
* Present dementia or neurological disorders which can increase cortical excitability
* Have psychotic or schizophrenic disorders
* Take drugs that reduce seizure threshold or spasticity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
American Spinal Injury Association Impairment Scale (ASIA), Assessment of change in motor scores from baseline to three weeks. | At baseline and after active intervention (i.e five consecutive days of rTMS) and sham (i.e five consecutive days of placebo rTMS). In a period of three weeks.
  The ASIA Motor Score is derived from part of the assessment for the International Standards for Neurological Classification of Spinal Cord Injury. It involves testing the strength of ten key muscles on each side of the body in the supine position (e.g., elbow flexors, wrist extensors, hip flexors, quadriceps, dorsiflexors) on a scale of 0 = no contraction to 5 = normal resistance through full range of motion. Scores are summed to give a total possible score of 50 for the upper extremities and 50 for the lower extremities.

SECONDARY OUTCOMES:
American Spinal Injury Association Impairment Scale (ASIA), Assessment of change in sensory scores from baseline to three weeks.sensory score. | At baseline and after active intervention (i.e five consecutive days of rTMS) and sham (i.e five consecutive days of placebo rTMS). In a period of three weeks.
  The ASIA Sensory score is also part of the assessment for the International Standard for Neurological Classification of Spinal Cord Injury. It involves testing pinprick and light touch sensation at key points representing each dermatome. Pin-prick and light-touch sensation of each dermatome is separately scored on a 3-point scale (0, 1 and 2). Scores will be summed to give a total possible score of 224 where a higher score indicates better sensation than a lower score.
Fugl-Meyer Scale for Upper and Lower Members, Assessment of change in motor scores from baseline to three weeks. | At baseline and after active intervention (i.e five consecutive days of rTMS) and sham (i.e five consecutive days of placebo rTMS). In a period of three weeks.
Electromyography (lower limbs), Assessment of change in motor function from baseline to three weeks. | At baseline and after active intervention (i.e five consecutive days of rTMS) and sham (i.e five consecutive days of placebo rTMS). In a period of three weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando H Magalhaes, Ph.D., Principal Investigator — University of Sao Paulo
Locations (1):
- Universidade Estadual da Paraiba, Campina Grande, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belci M, Catley M, Husain M, Frankel HL, Davey NJ. Magnetic brain stimulation can improve clinical outcome in incomplete spinal cord injured patients. Spinal Cord. 2004 Jul;42(7):417-9. doi: 10.1038/sj.sc.3101613. PMID 15111994
- [Background] Benito J, Kumru H, Murillo N, Costa U, Medina J, Tormos JM, Pascual-Leone A, Vidal J. Motor and gait improvement in patients with incomplete spinal cord injury induced by high-frequency repetitive transcranial magnetic stimulation. Top Spinal Cord Inj Rehabil. 2012 Spring;18(2):106-12. doi: 10.1310/sci1802-106. PMID 23459246
- [Background] Bunday KL, Perez MA. Motor recovery after spinal cord injury enhanced by strengthening corticospinal synaptic transmission. Curr Biol. 2012 Dec 18;22(24):2355-61. doi: 10.1016/j.cub.2012.10.046. Epub 2012 Nov 29. PMID 23200989
- [Background] Defrin R, Grunhaus L, Zamir D, Zeilig G. The effect of a series of repetitive transcranial magnetic stimulations of the motor cortex on central pain after spinal cord injury. Arch Phys Med Rehabil. 2007 Dec;88(12):1574-80. doi: 10.1016/j.apmr.2007.07.025. PMID 18047871
- [Background] Jette F, Cote I, Meziane HB, Mercier C. Effect of single-session repetitive transcranial magnetic stimulation applied over the hand versus leg motor area on pain after spinal cord injury. Neurorehabil Neural Repair. 2013 Sep;27(7):636-43. doi: 10.1177/1545968313484810. Epub 2013 Apr 11. PMID 23579183
- [Background] Kang BS, Shin HI, Bang MS. Effect of repetitive transcranial magnetic stimulation over the hand motor cortical area on central pain after spinal cord injury. Arch Phys Med Rehabil. 2009 Oct;90(10):1766-71. doi: 10.1016/j.apmr.2009.04.008. PMID 19801069
- [Background] Kumru H, Murillo N, Samso JV, Valls-Sole J, Edwards D, Pelayo R, Valero-Cabre A, Tormos JM, Pascual-Leone A. Reduction of spasticity with repetitive transcranial magnetic stimulation in patients with spinal cord injury. Neurorehabil Neural Repair. 2010 Jun;24(5):435-41. doi: 10.1177/1545968309356095. Epub 2010 Jan 6. PMID 20053952
- [Background] Kuppuswamy A, Balasubramaniam AV, Maksimovic R, Mathias CJ, Gall A, Craggs MD, Ellaway PH. Action of 5 Hz repetitive transcranial magnetic stimulation on sensory, motor and autonomic function in human spinal cord injury. Clin Neurophysiol. 2011 Dec;122(12):2452-61. doi: 10.1016/j.clinph.2011.04.022. Epub 2011 May 19. PMID 21600843
- [Background] Lammertse D, Tuszynski MH, Steeves JD, Curt A, Fawcett JW, Rask C, Ditunno JF, Fehlings MG, Guest JD, Ellaway PH, Kleitman N, Blight AR, Dobkin BH, Grossman R, Katoh H, Privat A, Kalichman M; International Campaign for Cures of Spinal Cord Injury Paralysis. Guidelines for the conduct of clinical trials for spinal cord injury as developed by the ICCP panel: clinical trial design. Spinal Cord. 2007 Mar;45(3):232-42. doi: 10.1038/sj.sc.3102010. Epub 2006 Dec 19. PMID 17179970
- [Background] Oudega M, Perez MA. Corticospinal reorganization after spinal cord injury. J Physiol. 2012 Aug 15;590(16):3647-63. doi: 10.1113/jphysiol.2012.233189. Epub 2012 May 14. PMID 22586214
- [Background] Tazoe T, Perez MA. Effects of repetitive transcranial magnetic stimulation on recovery of function after spinal cord injury. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S145-55. doi: 10.1016/j.apmr.2014.07.418. Epub 2014 Aug 29. PMID 25175159
- [Background] Yilmaz B, Kesikburun S, Yasar E, Tan AK. The effect of repetitive transcranial magnetic stimulation on refractory neuropathic pain in spinal cord injury. J Spinal Cord Med. 2014 Jul;37(4):397-400. doi: 10.1179/2045772313Y.0000000172. Epub 2013 Nov 11. PMID 24621025
- [Derived] de Araujo AVL, Barbosa VRN, Galdino GS, Fregni F, Massetti T, Fontes SL, de Oliveira Silva D, da Silva TD, Monteiro CBM, Tonks J, Magalhaes FH. Effects of high-frequency transcranial magnetic stimulation on functional performance in individuals with incomplete spinal cord injury: study protocol for a randomized controlled trial. Trials. 2017 Nov 6;18(1):522. doi: 10.1186/s13063-017-2280-1. PMID 29110687